CLINICAL TRIAL: NCT04629391
Title: Anatomic Versus Reverse Shoulder Arthroplasty for Primary Glenohumeral Osteoarthritis. a Randomized Prospective Study
Brief Title: Anatomic TSA Vs RTSA for Glenohumeral Arthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: La Tour Hospital (Other)
Responsible Party: Principal Investigator, Dr. Alexandre Lädermann, Principal Investigator, La Tour Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-02471
Record Dates: First submitted 2020-08-25; First posted 2020-11-16 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Arthritis Shoulder
Keywords: shoulder; primary osteoarthritis; Range of motion; clinical outcomes; radiographic outcomes; anatomic prosthesis; reverse prosthesis; Arthroplasty
MeSH Terms: interventions — Arthroplasty, Replacement, Shoulder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: While the patients and care providers will be aware of the type of prosthesis, the physicians who assessed the outcomes and analyzed the data will be blinded to this information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anatomic TSA (Active Comparator): The control group will receive through a deltopectoral approach an anatomic total shoulder arthroplasty (TSA) for a primary glenohumeral arthritis
  Interventions: Device: Total shoulder arthroplasty
- RTSA (Experimental): The experimental group will receive through a deltopectoral approach a reverse total shoulder arthroplasty RTSA for a primary glenohumeral arthritis
  Interventions: Device: Total shoulder arthroplasty

INTERVENTIONS:
Device: Total shoulder arthroplasty — A prosthesis (either anatomic or reverse) will be implanted in shoulders patients that suffer from primary glenohumeral arthritis.

SUMMARY:
There are no published prospective studies that compared 2-year functional outcomes of RTSA and anatomic TSA for the treatment of primary glenohumeral osteoarthritis with intact rotator cuffs and no excessive glenoid retroversion. The primary goal of our prospective randomized study is to determine whether RTSA have at least as good results as anatomic TSA (non-inferiority), in patients with glenohumeral osteoarthritis, without rotator cuff tears nor significant glenoid retroversion.

DETAILED DESCRIPTION:
Total anatomic shoulder arthroplasty (TSA) is an effective treatment of severe glenohumeral osteoarthritis, with significant improvement in shoulder pain and function. Concerns about glenoid loosening, associated with difficult revision procedures and disappointing outcomes, have however been raised.

Reverse total shoulder arthroplasty (RTSA) was designed with a medialized center of rotation to treat cuff tear arthropathy. Favorable early reports led to the expansion of primary indications of RTSA to proximal humeral fractures as well as osteoarthritis with poor glenoid bone stock. Recent reports revealed excellent clinical results of RTSA for primary glenohumeral arthropathy with intact rotator cuff and a low rate of complications.

Retrospective studies comparing functional results - of anatomic TSA for treating glenohumeral osteoarthritis with RTSA for rotator cuff arthropathy - found equivalent or greater improvements in American Shoulder and Elbow Surgeons score (ASES) at >2-year follow-up. In a study comparing anatomic TSA to RTSA for the treatment of glenohumeral osteoarthritis with intact rotator cuffs, Steen et al. reported equivalent functional results at >2-year follow-up. The retrospective matched cohort study could, however, not eliminate biases, such that RTSA patients had higher preoperative glenoid retroversion than anatomic TSA patients. The authors therefore hypothesize that, in patients treated for glenohumeral osteoarthritis without excessive glenoid retroversion, RTSA will render better functional outcomes than anatomic TSA, at 2 postoperative years. Many other studies confirmed in 2019 Steen's hypothesis. Moreover, several studies revealed good long-term survivorship after RTSA.

There are no published prospective studies that compared 2-year functional outcomes of RTSA and anatomic TSA for the treatment of primary glenohumeral osteoarthritis with intact rotator cuffs and no excessive glenoid retroversion. The primary goal of our prospective randomized study is to determine whether RTSA have at least as good results as anatomic TSA (non-inferiority), in patients with glenohumeral osteoarthritis, without rotator cuff tears nor significant glenoid retroversion.The secondary goals are 1) to evaluate whether RTSA eventually grants superior postoperative clinical and radiographic outcomes than anatomic TSA (superiority), 2) to determine whether RTSA is associated with fewer postoperative complications than anatomic TSA.

ELIGIBILITY:
Inclusion Criteria:

* Primary glenohumeral arthritis,
* Intact rotator cuff,
* No important glenoid bone loss (cf exclusion criteria),
* Patients between 65 and 85 years old
* Informed Consent as documented by signature (Appendix Informed Consent Form).

Exclusion Criteria:

* B2 glenoid with > 80% posterior humeral head subluxation or greater 25 degrees neoglenoid retroversion,
* B3 and C type glenoids,
* Full thickness rotator cuff tear,
* Acute or malunited proximal humeral fracture,
* Chronic locked dislocation
* Rheumatoid arthritis,
* Revision surgery or surgical antecedents,
* Tumors,
* Axillary nerve damage,
* Non-functioning deltoid muscle,
* Glenoid vault deficiency precluding baseplate fixation,
* Infection and neuropathic joints,
* Known or suspected non-compliance, drug or alcohol abuse,
* Patients incapable of judgement or under tutelage,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, contraindication for CT scan etc. of the participant,
* Enrolment of the investigator, his/her family members, employees and other dependent persons.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 296 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in American Shoulder and Elbow Surgeons score (ASES) | Between baseline and 2 postoperative years
  General clinical score (0-100, with 100 being the best score possible)

SECONDARY OUTCOMES:
Change in Subjective Shoulder Value (SSV) | Between baseline and 2 postoperative years
  General clinical score (0-100, with 100 being the best score possible)
Change in Range of motion in degrees | Between baseline and 2 postoperative years
  (anterior forward flexion, external rotation at the side, internal rotation to nearest spinal level)
Complication rates | 2 postoperative years.
Change in pain on visual analogic scale (pVAS) | Between baseline and 2 postoperative years
  General clinical score (0-10, with 10 the worst score possible)
Change in Constant score | Between baseline and 2 postoperative years
  General clinical score (0-100, with 100 being the best score possible)
Change in Short Form -12 (SF-12) | Between baseline and 2 postoperative years
  General clinical score (0-100, with 100 being the best score possible)
Radiographic outcomes | 2 postoperative years
  Rates of aseptic loosening, implant migration, implant tilt, scapular notching, glenoid bone loss as defined previously by the investigator

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Lädermann, MD, Principal Investigator — La Tour Hospital
Locations (1):
- La Tour Hospital, Meyrin, Switzerland

IPD SHARING:
Plan to Share IPD: No